CLINICAL TRIAL: NCT05968976
Title: The TREMBLE Study: Multicentre Randomized Controlled Trial of Awake Versus Asleep Tractography Based Deep Brain Stimulation for Essential Tremor
Brief Title: Multicentre RCT of Awake Versus Asleep Tractography Based DBS for ET
Acronym: TREMBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University Medical Center Groningen (Other); Medical Center Haaglanden (Other); The Elisabeth-TweeSteden Hospital (Other); Maastricht University Medical Center (Other); Radboud University Medical Center (Other); Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, Maarten Bot, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL80368.018.23
Record Dates: First submitted 2023-06-09; First posted 2023-08-01 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor; Deep Brain Stimulation; Diffusion Tensor Imaging; Magnetic Resonance; Central Nervous System Diseases
MeSH Terms: conditions — Essential Tremor; Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: The study will be a multicentre prospective randomized open label blinded (PROBE) endpoint trial comparing thalamic DBS under general versus local anesthesia
Who Masked: Outcomes Assessor
Masking Description: Because both patient and neurosurgeon are aware of receiving general or local anesthesia, it is not possible to blind them for treatment assignment. Patients will be instructed not to reveal the received treatment with the physician performing the 6-month assessments and neuropsychological evaluation in order to secure a blinded end-point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 55 patients with essential tremor receive awake DBS (Active Comparator)
  Interventions: Procedure: Awake DBS
- 55 patients with essential tremor receive asleep DBS (Experimental)
  Interventions: Procedure: Asleep DBS

INTERVENTIONS:
Procedure: Awake DBS — 55 patients receive awake DBS (current standard procedure)
  Arms: 55 patients with essential tremor receive awake DBS
Procedure: Asleep DBS — 55 patients receive asleep DBS
  Arms: 55 patients with essential tremor receive asleep DBS

SUMMARY:
Rationale: Deep brain stimulation (DBS) of the thalamus is an effective surgical treatment for patients with disabling essential tremor, despite optimal pharmacological treatment. To date, the standard DBS procedure is performed under local anesthesia which is very burdensome for patients. It is now possible to directly visualize the target (motor) area in the thalamus due to advances in modern imaging techniques. DBS surgery could be performed under general anesthesia (asleep).

Objective: The primary objective of the study is to determine whether asleep thalamic DBS surgery provides an equal tremor reduction compared to awake thalamic DBS surgery, measured by the clinically validated Essential Tremor Rating Assessment Scale after six months of DBS.

Secondary outcomes are: disease related daily functioning, adverse effects, operation time, quality of life, patient satisfaction with treatment outcome and patient evaluation of treatment burden.

Study design: The study will be a multicentre prospective randomized open label blinded (PROBE) endpoint trial comparing thalamic DBS under general versus local anesthesia.

Study population: A total of 110 patients with disabling essential tremor despite optimal pharmacological treatment will be randomized.

Intervention (if applicable): Patients will be randomized for asleep DBS or awake DBS. According to the standard DBS procedure, two brain-electrodes are connected to an implanted neurostimulator, which is placed subcutaneously in the subclavicular area

Main study parameter/endpoints: The primary outcome measure is the change in tremor score on the Essential Tremor Rating Assessment Scale after 6 months of thalamic DBS.

The secondary outcome measures are the Amsterdam Linear Disability Score for functional health status, Quality of Life in Essential Tremor Questionnaire, patient satisfaction with the treatment, patient evaluation of treatment burden, operating time, hospitalization time, change of tremor medication, side effects and complications.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Awake DBS at present is very burdensome and by many patients and health care providers considered to be an overly invasive treatment for essential tremor. Through this trial, we aim to investigate whether asleep DBS in essential tremor can become the new treatment standard. This is expected to increase the accessibility for DBS and subsequently would allow more people with essential tremor to be helped, as well as in an earlier stage of their disease than currently; more patients will benefit for a longer time period from DBS. Asleep DBS will have a shorter procedure length. The proposed research project involves treatment options that are standard care in daily practice. The therapies will not be combined with other research products. Both treatments have a low risk of serious complications and a higher risk of minor side effects. Regular follow up will be used. Participation in this study constitutes moderate risk according to NFU criteria for human research.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Essential tremor Essential tremor is the most common neurological movement disorder and often begins at an early age. In 20 to 30 years, the disorder develops to an advanced stage, in which patients are severely disabled by the tremor (trembling, shaking) of their hands in particular (and additional shaking of the head, legs and vocal cords may occur). In most severe cases, drug treatment only partially suppresses the tremor, and also loses effect over time. As a result, patients can no longer use their hands properly, for example, when eating and carrying out their activities of daily living. Patients become care-dependent. In addition, the involuntary tremor is socially disruptive and prevents patients from showing up in public places; they become socially isolated.

Because the tremor increases gradually in severity (over decades), patients and their immediate environment adapt their lives accordingly. For example, they drink with a straw, eat foods that are easy to scoop up and avoid social occasions because the trembling is perceived as disturbing. Often the possibility of treatment with DBS could have been considered years earlier, however this possibility is unknown to both patient and caregiver, or the DBS is seen as experimental.

Thalamic DBS is an effective surgical treatment for patients with disabling essential tremor who have severe limitations in their functioning despite pharmacological treatment. During the surgical placement of DBS brain electrodes, patients are awake so that the effect of the electrode implantation can be monitored. Awake DBS surgery is extremely burdensome and therefore prevents many patients from undergoing the treatment. To increase accessibility to DBS, we want to perform the surgery asleep.

Functional stereotactic neurosurgery Currently the standard DBS procedure is performed awake. Patients need to be awake during the surgery as the optimal placement of the stimulation electrodes into the brain is confirmed by intra-operative clinical testing. This procedure is extremely burdensome for patients: 1) cranial injections are needed for local anesthesia 2) a frame is fixed to their head with four bone-pins 3) they are secured to the operating table for the procedure 4) burr holes are drilled into their skull and 5) electrodes are implanted during which patients are hours continuously tested for DBS effect.

Due to advances in MRI tractography techniques (displaying connecting pathways between brain regions using magnetic resonance imaging) the target area for DBS can now be clearly visualized and therefore it may be possible to perform the entire procedure asleep without the need for intraoperative clinical testing. Several studies, including a recent randomized controlled DBS trial in Parkinson's disease at the Amsterdam UMC, have shown that asleep DBS is safe. This trial also showed that Parkinson's patients experienced asleep DBS as less invasive, both psychologically and physically. Logically, asleep DBS also lowers the burden of surgery for essential tremor patients. This is expected to increase the accessibility for DBS. This would allow more people with essential tremor to be helped, as well as in an earlier stage of their disease; more patients will benefit for a longer time period from DBS. To determine whether asleep DBS for essential tremor suppresses tremor as well as awake DBS, a comparative study is warranted.

General anesthesia General anesthesia is routinely used in different types of surgery. In the Amsterdam UMC, all Parkinson's disease patients, patients with dystonia, obsessive-compulsive disorder, anorexia or epilepsia, where peri-operative testing is not necessary, the electrodes are placed asleep. The patients receiving electrode insertion under local anesthesia will receive general anesthesia to implant the pulse generator subcutaneously. The procedure is described in chapter 4- Treatment of subjects.

Asleep compared to awake thalamic DBS for essential tremor

Tremor suppression Since the 1980s, DBS for essential tremor was targeting the thalamus, a deep-seated grey matter brain nucleus. Current emphasis in the field of DBS is on neural networks rather than separate nuclei in the brain. Several studies showed essential tremor to arise from pathological network activity in cerebellar-cortical projections. In recent years the MRI techniques for visualisation of brain networks became widely available in DBS software modules. The 3-Tesla MRI diffusion deterministic tractography is a powerful tool to visualise structural connections between brain nuclei and different cortical areas. In recent years several DBS groups reported about using tractography to visualize the cerebellar-cortical projections, or dentato-rubro-thalamic-tract (DRT), in DBS for essential tremor. By visualizing the DRT, a direct target for DBS electrode placement was generated. In the Amsterdam UMC, we have been evaluating DRT for DBS in essential tremor from 2017. Since then, we published two major studies evaluating DRT based DBS in essential tremor. First, we studied the optimization of deterministic DRT tractography by applying a standardized technique for constructing the tract and using a newly developed MRI sequence; the fast grey matter acquisition T1 inversion recovery (FGATIR). This enabled us to construct an approximation of the DRT that strongly correlated with optimal tremor control for DBS. In the following prospective clinical study we implemented this DRT technique for all our DBS cases in essential tremor. We showed that during intraoperative testing the pre-determined trajectory based on DRT depiction showed complete tremor suppression in all cases. Intraoperative testing confirmed the optimal location for tremor suppression was accurately indicated by the (preoperative generated) DRT. These two studies show DRT based DBS provides a direct target area for DBS in essential tremor and possibly omits the need for intraoperative, awake, testing.

Adverse effects Several studies, including a recent randomized controlled DBS trial in Parkinson's disease at the Amsterdam UMC, have shown that asleep DBS is safe. This trial also showed that people experience asleep DBS less invasive, both psychologically and physically.6 Multiple studies report on dysarthria and gait ataxia after thalamic/DRT DBS in essential tremor. When dysarthria occurs during awake test stimulation, it is usually not possible to differentiate between effects of intraoperative testing and edema due to electrode introduction. Moreover, in a third of patients stimulation-induced dysarthria during follow up was not preceded by dysarthria during test stimulation, indicating that this is not a reliable predictor for chronic effects. Gait ataxia cannot be tested during surgery, and usually occurs gradually during follow up, both with or without pre-existing balance difficulties. This shows awake intraoperative testing cannot be used to prevent these side effects from occurring during follow up. Another known side effect can be induced by co-stimulation of the corticospinal fibres, which are located (passing) near the thalamus. In our recent essential tremor studies we have shown that tractography can also be used to visualize the corticospinal fibres, ensuring sufficient distance to the DBS electrode trajectory for preventing co-stimulation (which would result in involuntary muscle contractions).

In sum, due to advancing insights in essential tremor pathophysiology and MRI tractography techniques, it is now possible to directly visualize part of the brain tremor network involved in the occurrence of tremor, the dentato-rubro-thalamic-tract. In awake DBS, this tract provided a direct target and showed high correlation with optimal tremor control, with a comparable side effect profile. DBS surgery could therefore now be performed asleep. To our knowledge, no randomized controlled trial has been done to compare the outcome between awake and asleep tractography guided DBS in essential tremor.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Idiopathic essential tremor
* Disabling tremor despite optimal pharmacological treatment
* A life expectancy of at least two years

Exclusion Criteria:

* Legally incompetent adults;
* Previous tremor-neurosurgery (e.g., DBS, thalamotomy);
* Contraindications for DBS surgery, such as a physical disorder making surgery hazardous;
* Psychosis;
* Current depression;
* Unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Essential Tremor Rating Assessment Scale (TETRAS) | assessment will be done before DBS and after 6 months of DBS
  The amount of decrease in motor symptoms indicated by change in the disease-specific Essential Tremor Rating Assessment Scale (TETRAS) after six months of deep brain stimulation. The TETRAS scores are between 0 and 64; higher scores indicating worse (more severe) tremor symptoms.

SECONDARY OUTCOMES:
The Amsterdam Linear Disability Score for functional health status | assessment will be done before DBS and after 6 months of DBS
  The Amsterdam Linear Disability Score (ALDS) is a generic itembank which measures disability, as expressed by the ability to perform activities of daily living. These scores are linearly transformed into values between 0 and 100. Lower scores indicate more disability.
Quality of Life in Essential Tremor Questionnaire | assessment will be done before DBS and after 6 months of DBS
  The Quality of Life in Essential Tremor Questionnaire (QUEST) is a 30-item scale developed specifically for patients with essential tremor to measure items impacting perceived quality of life (QOL) that generic QOL measures do not effectively capture, including activities of daily living that are affected by essential tremor. The QUEST was made to be relatively brief and easy for patients to use.
Global Impression of Change | assessment will be done before DBS and after 6 months of DBS
  The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. The CGI actually comprises two companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale.
EQ-5D-5L | assessment will be done before DBS and after 6 months of DBS
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 2024

REFERENCES:
- [Background] 1. Song P, Zhang Y, Zha M, et al. The global prevalence of essential tremor, with emphasis on age and sex: A meta-analysis. J Glob Health. Apr 10 2021;11:04028. 2. Schuurman PR, Bosch DA, Merkus MP, Speelman JD. Long-term follow-up of thalamic stimulation versus thalamotomy for tremor suppression. Movement disorders : official journal of the Movement Disorder Society. Jun 15 2008;23(8):1146-1153. 3. Bot M, van Rootselaar F, Contarino MF, et al. Deep Brain Stimulation for Essential Tremor: Aligning Thalamic and Posterior Subthalamic Targets in 1 Surgical Trajectory. Oper Neurosurg (Hagerstown). Aug 1 2018;15(2):144-152. 4. Bot M, van Rootselaari AF, Odekerken V, et al. Evaluating and Optimizing Dentato-Rubro-Thalamic-Tract Deterministic Tractography in Deep Brain Stimulation for Essential Tremor. Oper Neurosurg (Hagerstown). Sep 25 2021. 5. Bot M, Pauwels R, van den Munckhof P, et al. The Fast Gray Matter Acquisition T1 Inversion Recovery Sequence in Deep Brain Stimulation: Introducing the Rubral Wing for Dentato-Rubro-Thalamic Tract Depiction and Tremor Control. Neuromodulation. Jan 15 2022. 6. Holewijn RA, Verbaan D, van den Munckhof PM, et al. General Anesthesia vs Local Anesthesia in Microelectrode Recording-Guided Deep-Brain Stimulation for Parkinson Disease: The GALAXY Randomized Clinical Trial. JAMA Neurol. Sep 7 2021. 7. Graat I, Mocking RJT, Liebrand LC, et al. Tractography-based versus anatomical landmark-based targeting in vALIC deep brain stimulation for refractory obsessive-compulsive disorder. Mol Psychiatry. Dec 2022;27(12):5206-5212. 8. Nowacki A, Barlatey S, Al-Fatly B, et al. Probabilistic Mapping Reveals Optimal Stimulation Site in Essential Tremor. Ann Neurol. May 2022;91(5):602-612. 9. Coenen VA, Sajonz B, Prokop T, et al. The dentato-rubro-thalamic tract as the potential common deep brain stimulation target for tremor of various origin: an observational case series. Acta neurochirurgica. May 2020;162(5):1053-1066. 10. Akram H, Dayal V, Mahlknecht P, et al. Connectivity derived thalamic segmentation in deep brain stimulation for tremor. Neuroimage Clin. 2018;18:130-142. 11. Nowacki A, Schlaier J, Debove I, Pollo C. Validation of diffusion tensor imaging tractography to visualize the dentatorubrothalamic tract for surgical planning. Journal of neurosurgery. Mar 23 2018;130(1):99-108. 12. Coenen VA, Allert N, Paus S, Kronenburger M, Urbach H, Madler B. Modulation of the Cerebello-Thalamo-Cortical Network in Thalamic Deep Brain Stimulation for Tremor: A Diffusion Tensor Imaging Study. Neurosurgery. Dec 2014;75(6):657-669. 13. Kremer NI, Pauwels RWJ, Pozzi NG, et al. Deep Brain Stimulation for Tremor: Update on Long-Term Outcomes, Target Considerations and Future Directions. J Clin Med. Aug 5 2021;10(16).